CLINICAL TRIAL: NCT04619888
Title: Follow-up of Heart Failure Patients with an Implantable Cardiac Defibrillator Enabled with the HeartLogic Algorithm - HeartLogic France Study
Brief Title: HeartLogic France Study: Heart Failure Patients Managed with the HeartLogic Algorithm
Status: Completed | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: HeartLogic France Study
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure
Keywords: Implantable cardioverter defibrillator; quality of life
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — 1 dry tube, 1 EDTA tube and 1 lithium heparin tube
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- HeartLogic cohort: Patients implanted with a defibrillator enabling HeartLogic
  Interventions: Diagnostic Test: HeartLogic

INTERVENTIONS:
Diagnostic Test: HeartLogic — In case of HeartLogic index ≥16, the investigator will contact the patient to assess the patient's clinical condition and possibly adjust the heart failure treatment. The management will be standardized across centers according to the Manage-HF protocol.

SUMMARY:
Heart Failure (HF) is a chronic disease that leads to numerous rehospitalisations and affects more than one million people in France.

The main objective of this prospective multicentric French study is to describe the annual rate of unplanned hospitalisations for heart failure in a cohort of patients managed by a HeartLogic algorithm.

Patients will be included if they fulfill the following requirements 1/Patient implanted with a cardiac defibrillator with or without resynchronisation with the HeartLogic index (RESONATE family, Boston Scientific); 2/History of heart failure (left ventricular ejection fraction ≤40 %; or at least one episode of clinical heart failure with elevated NT pro BNP≥450 ng/L).

If a HeartLogic index ≥16 is noticed, the investigator will contact the patient to assess the patient's clinical condition and possibly adjust the heart failure treatment.

DETAILED DESCRIPTION:
Heart Failure (HF) is a chronic disease that leads to numerous rehospitalisations and affects more than one million people in France.

The main objective of this prospective multicentric French study is to describe the annual rate of unplanned hospitalisations for heart failure in a cohort of patients managed by a HeartLogic algorithm.

310 patients will be included if they fulfill the following requirements 1/Patient implanted with a cardiac defibrillator with or without resynchronisation with the HeartLogic index (RESONATE family, Boston Scientific); 2/History of heart failure (left ventricular ejection fraction ≤40 %; or at least one episode of clinical heart failure with elevated NT pro BNP≥450 ng/L).

The HeartLogic index will be monitored remotely on a weekly basis for 12 months and in case of HeartLogic index ≥16, the local investigator will contact the patient for assessment and adjust HF treatment as necessary. The primary endpoint is unscheduled hospitalization for HF. A blind and independent committee will adjudicate the events. Blood samples will be collected for biobanking, and quality of life will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Patient implanted with a cardiac defibrillator, with or without resynchronization, enabled with the HeartLogic index (RESONATE family, Boston Scientific)
* History of heart failure (left ventricular ejection fraction ≤40 %; or at least one episode of clinical heart failure with elevated NT pro BNP≥450 ng/L)

Exclusion Criteria:

* Concomitant presence of a heart failure device other than cardiac resynchronisation such as a left ventricular assist device or a device for modulating cardiac contractility.
* Heart transplant project, or heart transplant patient
* Glomerular filtration rate <30 ml/mn/m2 or dialysis,
* Life expectancy ≤ 6 months
* Remote monitoring of HeartLogic is not possible.
* Refusal to take medication for heart failure
* Patient with a mechanical heart valve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart failure patients equipped with an ICD
Sampling Method: Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Hospitalisation for heart failure | During 12 months
  Annual rate of unplanned hospitalisations for heart failure

SECONDARY OUTCOMES:
Cardiovascular mortality | During 12 months
  Annual cardiovascular mortality rate
Heart failure related mortality | During 12 months
  Annual death rate from heart failure
Unplanned hospitalisation due to ventricular arrhythmia | During 12 months
  Annual rate of unplanned hospitalisation due to ventricular arrhythmia
Unplanned hospitalisations due to atrial arrhythmia | During 12 months
  Annual rate of unplanned hospitalisations due to atrial arrhythmia
Hospitalisation duration related to heart failure, ventricular or atrial arrhythmia | During 12 months
  Annual rate of hospitalisation days related to heart failure, ventricular or atrial arrhythmia
Patient quality of life using the Kansas City Cardiomyopathy Questionnaire | At baseline and 1 year
  Scale title : KCCQ; Score between 0 and 100; higher scores reflect better health status
Evolution of the average HeartLogic index each week over a 12-month period | During 12 months
  Scale title HL index; The lower value is 0 and there is no upper limit; A higher value reflects a higher probability of heart failure
Effect of iSGLT2 on HeartLogic index, atrial arrhythmias and ventricular arrhythmias | During 12 months
  Describe HeartLogic index, atrial arrhythmias and ventricular arrhythmias before and after iSGLT2 medication initiation and between patient treated or not treated with iSGLT2 treatment
Safety of preemptive congestion treatment based on HeartLogic index | During 12 months
  Combined "diuretic intolerance" criteria comprising either an increase in creatinine ≥30%, or an increase or decrease in kaliemia≥30%, or a decrease in natremia ≥30% between the time of the HeartLogic alert and the end of diuretic treatment, or the occurrence of symptomatic hypotension secondary to the initiation or increase in diuretic treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigue Garcia, Study Director — University Hospital of Poitiers
Locations (10):
- France (10):
  - University hospital of Brest, Brest
  - University hospital of Grenoble, Grenoble
  - Hospital of Lorient, Lorient
  - Clinique du Confluent, Nantes
  - University Hospital of Nantes, Nantes
  - Hopital Europeen G Pompidou, Paris
  - Hopital La Salpétrière, Paris
  - University Hospital of Poitiers, Poitiers
  - Clinique Pasteur, Toulouse
  - University Hospital of Tours, Tours

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Garcia R, Gras D, Mansourati J, Defaye P, Bisson A, Boveda S, Durocher L, Gandjbakhch E, Gras M, Gueffet JP, Himbert C, Jacon P, Khattar P, Lequeux B, Li A, Mansourati V, Minois D, Marijon E, Pierre B, Ragot S, Probst V, Degand B. Impact and safety of remote monitoring of heart failure patients managed with the HeartLogic algorithm: the HeartLogic France Cohort Study. Eur Heart J Digit Health. 2025 Nov 13;7(2):ztaf133. doi: 10.1093/ehjdh/ztaf133. eCollection 2026 Mar. PMID 41624570